CLINICAL TRIAL: NCT01221363
Title: Reduction of Sitting Time - a Randomized Controlled Intervention Study
Brief Title: Reduction of Sitting Time: Sedentarism Intervention Trial
Acronym: SIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Lundbeck Foundation (Other); Sygekassernes Helsefond (Other)
Responsible Party: Principal Investigator, Allan Linneberg, Researchmanager, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCT00289237
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Results first posted 2015-01-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Life Style; Physical Activity; Sedentary Behavior
Keywords: Life style disease; Obesity; Sedentary behaviour; Cardiovascular biomarkers
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counselling (Active Comparator): Theory based individually tailored lifestyle counselling aimed at reduction of sitting time during leisure time and at work. Four individual sessions over a six months period.
  Interventions: Behavioral: Life style intervention
- Control group (No Intervention): No intervention control group

INTERVENTIONS:
Behavioral: Life style intervention — Reduction of sedentary behavior through theory-based individually tailored lifestyle intervention.
  Other Names: Life style counselling
  Arms: Lifestyle counselling

SUMMARY:
Recent studies have suggested that prolonged daily sitting time may in itself have a negative effect on health, even in people who engage in daily physical activity.

The aim of the present study is to explore whether individually tailored lifestyle counselling aimed at reducing TV-viewing and other sedentary activities during leisure time and at work, can reduce sitting time and waist circumference, weight and blood pressure; and improve serum lipid levels. From a population-based health survey, 150 adult men and women with more than 3.5 hours of daily leisure time sitting time are recruited and randomly assigned to 1) an intervention group or 2) a control group. The intervention group will participate in 4 individually tailored lifestyle intervention sessions focussing on reduction of daily sitting time. The control group will receive no intervention.

DETAILED DESCRIPTION:
Evidence for the health benefits of regular physical activity is clear and unanimous. Recently, observational studies have found that prolonged bouts of sitting time are associated with chronic disease and mortality, even in individuals who engage in regular physical activity. These new findings indicate that sedentary behaviour should be regarded as a distinct class of behaviour with independent effects on disease risk, separate from the behaviour of leisure time physical activity. Prolonged daily sitting time is prevalent in modern, western society, making further exploration into this field of research a relevant public health issue.

It remains to be tested, whether it is possible to reduce sedentary leisure time in adults and whether a reduction of sedentary leisure time will lead to a decrease in biological CVD risk factors.

The investigators hypothesize that sedentary behaviour during leisure time and at work may be reduced through a theory-based individually tailored lifestyle intervention.

Aim: To examine whether an individually tailored lifestyle intervention aimed at reducing TV-viewing and other sedentary activities during leisure time and at work, can reduce sitting time, waist circumference, BMI and blood pressure; and improve serum lipid level.

Study population: From the "Health2010" study, that was initiated February 2010 at the RCPH, 150 sedentary participants will be consecutively invited and randomised by computer-generated random numbers into A) an intervention group (n=75) and B) a control group (n=75), when visiting the RCPH for the health examination. The entire Health2010 population will comprise 4.000 men and women between 19 and 69 years of age.

Control group: The control group will be instructed to maintain their usual lifestyle, including physical activity level and sedentary behaviour. After the intervention period is terminated, participants in the control group will be given the written material (booklets etc.).

Primary outcome measure: Time engaging in sedentary activities (hours & minutes per day), as measured by ActivPAL. Secondary outcome measures: self-reported physical activity and sitting time, total cholesterol, HDL, triglycerides, LDL, weight, waist circumference, systolic and diastolic blood pressure. Outcome measures will be obtained at baseline (inclusion) and after 6 months.

A possible effect of the intervention on self-reported sedentary leisure time (primary outcome) and biological CVD risk factors (secondary outcomes) will be explored by comparison of intervention and control group at baseline and follow-up. Regression analysis and intention-to-treat analysis will be applied and a significance level of 0.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Minimum selfreported 3 ½ hours of sedentary leisure time per day

Exclusion Criteria:

* More than 8 hours of vigorous activity per week
* Physical handicap or illness that prevent reduction of sitting time
* Must be able to read and understand Danish

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torben Jørgensen, Prof. DrMedSc, Study Director — Research Centre for Prevention and Health, the Capital Region of Denmark
Locations (1):
- Research Centre for Prevention and Health, The Capital Region of Denmark, Glostrup Municipality, Denmark

REFERENCES:
- [Background] Otten JJ, Jones KE, Littenberg B, Harvey-Berino J. Effects of television viewing reduction on energy intake and expenditure in overweight and obese adults: a randomized controlled trial. Arch Intern Med. 2009 Dec 14;169(22):2109-15. doi: 10.1001/archinternmed.2009.430. PMID 20008695
- [Background] Dunstan DW, Barr EL, Healy GN, Salmon J, Shaw JE, Balkau B, Magliano DJ, Cameron AJ, Zimmet PZ, Owen N. Television viewing time and mortality: the Australian Diabetes, Obesity and Lifestyle Study (AusDiab). Circulation. 2010 Jan 26;121(3):384-91. doi: 10.1161/CIRCULATIONAHA.109.894824. Epub 2010 Jan 11. PMID 20065160
- [Background] Wijndaele K, Healy GN, Dunstan DW, Barnett AG, Salmon J, Shaw JE, Zimmet PZ, Owen N. Increased cardiometabolic risk is associated with increased TV viewing time. Med Sci Sports Exerc. 2010 Aug;42(8):1511-8. doi: 10.1249/MSS.0b013e3181d322ac. PMID 20139784
- [Background] Wijndaele K, Brage S, Besson H, Khaw KT, Sharp SJ, Luben R, Wareham NJ, Ekelund U. Television viewing time independently predicts all-cause and cardiovascular mortality: the EPIC Norfolk study. Int J Epidemiol. 2011 Feb;40(1):150-9. doi: 10.1093/ije/dyq105. Epub 2010 Jun 23. PMID 20576628
- [Background] Hamilton MT, Hamilton DG, Zderic TW. Role of low energy expenditure and sitting in obesity, metabolic syndrome, type 2 diabetes, and cardiovascular disease. Diabetes. 2007 Nov;56(11):2655-67. doi: 10.2337/db07-0882. Epub 2007 Sep 7. PMID 17827399
- [Background] Katzmarzyk PT, Church TS, Craig CL, Bouchard C. Sitting time and mortality from all causes, cardiovascular disease, and cancer. Med Sci Sports Exerc. 2009 May;41(5):998-1005. doi: 10.1249/MSS.0b013e3181930355. PMID 19346988
- [Background] Aadahl M, Kjaer M, Jorgensen T. Influence of time spent on TV viewing and vigorous intensity physical activity on cardiovascular biomarkers. The Inter 99 study. Eur J Cardiovasc Prev Rehabil. 2007 Oct;14(5):660-5. doi: 10.1097/HJR.0b013e3280c284c5. PMID 17925625
- See also: Research Centre for Prevention and Health, The Capital Region of Denmark — http://www.rcph.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 171 participants were consecutively included. However 5 patients withdrew before randomisation, leaving 166 participants to be included and randomised to either the intervention or the control group.
  Reasons for withdrawal were: 4 participants changed their mind because of lack of time, 1 participant reported skin reaction to monitor attachment.
Period: Overall Study
Arm/Group | Lifestyle Counselling | Control Group
Started | 93 | 73
Completed | 81 | 68
Not Completed | 12 | 5
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Counselling | Control Group | Total
Number analyzed (Participants) | 93 | 73 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (13.8) | 51.8 (14.3) | 52 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 36 | 95
  Male | 34 | 37 | 71
Region of Enrollment [Number; unit: participants]
  Denmark | 93 | 73 | 166

OUTCOME MEASURES:

1. Primary Outcome: Change in Objectively Measured Sitting Time From Baseline to 6 Months Follow-up
Description: Participants wore an ActivePAL monitor for seven days at inclusion and seven days at follow-up. The ActivePAL measures sitting time.
  Change in sitting time from baseline to 6 months follow up was evaluated.
Time Frame: 7 days of measurement / change in sitting time from baseline and 6 months follow-up
Population: Within group difference
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | Lifestyle Counselling | Control Group
Number analyzed (Participants) | 81 | 68
Hours per day | -0.27 (1.7) | 0.06 (1.7)

2. Secondary Outcome: Change in High Density Lipoprotein (HDL) From Baseline to 6 Months Follow-up.
Description: Blood samples are drawn at inclusion and at 6 months follow-up. Change in measured HDL (mmol/L) from baseline to 6 months follow-up
Time Frame: Change in measured HDL from baseline and 6 months follow-up
Measure: Mean (Standard Deviation); unit: mmol/Liter
Arm/Group | Lifestyle Counselling | Control Group
Number analyzed (Participants) | 81 | 68
mmol/Liter | -0.03 (0.2) | -0.02 (0.2)

ADVERSE EVENTS:
Time Frame: November 2010 to March 2012
Arm/Group | Lifestyle Counselling | Control Group
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/73
Other Adverse Events (participants affected / at risk) | 0/93 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No